CLINICAL TRIAL: NCT00111644
Title: A Randomized, Double-blind Study of the Effect of Beta-lactam on Treatment Response in Patients Hospitalized With Bacterial Pneumonia
Brief Title: A Study to Assess Beta-Lactam in the Treatment of Hospitalized Patients With Bacterial Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WI18273
Record Dates: First submitted 2005-05-24; First posted 2005-05-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Pneumonia, Bacterial
MeSH Terms: conditions — Pneumonia, Bacterial | interventions — Ceftriaxone; beta-Lactams

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: beta-lactam
- 2 (Experimental)
  Interventions: Drug: beta-lactam
- 3 (Active Comparator)
  Interventions: Drug: Ceftriaxone

INTERVENTIONS:
Drug: Ceftriaxone — 1000mg iv daily
  Arms: 3
Drug: beta-lactam — 750mg iv q 23h for 3-14 days
  Arms: 1
Drug: beta-lactam — 1500mg iv q 12h for 3-14 days
  Arms: 2

SUMMARY:
This study will assess the efficacy and safety of intravenous beta-lactam, in comparison with ceftriaxone, in hospitalized patients with community-acquired pneumonia not caused by Legionella. The anticipated time on study treatment is 3-12 months and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients at least 18 years of age;
* hospitalization with community-acquired pneumonia or development of pneumonia within 48 hours of being hospitalized for another reason;
* fever;
* new or increased productive cough;
* chest pain, shortness of breath, or rapid breathing.

Exclusion Criteria:

* requiring intubation or ventilation;
* nursing home or extended care within 60 days before study;
* concomitant bacterial infection requiring antibiotics;
* long-term immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2005-03; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Clinical cure rate\n\n | End of study visit (7-10 days after end of treatment)

SECONDARY OUTCOMES:
Adverse events, vital signs, laboratory parameters\n | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- United States (6):
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Detroit, Michigan
  - Butte, Montana
  - Holmdel, New Jersey
  - Winston-Salem, North Carolina
- Argentina (6):
  - Buenos Aires
  - Ciudadela
  - Córdoba
  - Granadero Baigorria
  - Paraná
  - Rosario
- Bulgaria (2):
  - Rousse
  - Sofia
- Chile (2):
  - Santiago
  - Valdivia
- Zagreb, Croatia
- Hungary (4):
  - Budapest
  - Nyíregyháza
  - Törökbálint
  - Zalaegerszeg
- Latvia (2):
  - Daugavpils
  - Riga
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Lima, Peru
- Romania (3):
  - Bucharest
  - Constanța
  - Craiova
- Slovakia (3):
  - Banská Bystrica
  - Nitra
  - Poprad